CLINICAL TRIAL: NCT00218387
Title: CBT and Modafinil for Cocaine Addiction
Brief Title: Modafinil Combined With Cognitive Behavior Therapy to Treat Cocaine Addiction - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Robert Malcolm, Professor of Psychiatry, Family Medicine & Pediatrics, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-16368-1; R01DA016368 (NIH); R01-16368-1; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-03

CONDITIONS: Cocaine Dependence
Keywords: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 200mg Modafinil (Experimental): 200mg Modafinil
  Interventions: Drug: Modafinil
- 400mg Modafinil (Experimental): 400mg Modafinil
  Interventions: Drug: Modafinil
- Matching Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Modafinil — 200mg Modafinil
  Other Names: Provigil
  Arms: 200mg Modafinil
Drug: Modafinil — 400mg Modafinil
  Other Names: Provigil
  Arms: 400mg Modafinil
Drug: Matching Placebo — Matching Placebo
  Arms: Matching Placebo

SUMMARY:
Cocaine addiction is a serious health problem with no available medical treatment for preventing relapse. Modafinil, a medication that enhances mood, increases energy, and improves concentration, may be useful in preventing relapse among individuals with cocaine addiction. This study will evaluate the effectiveness of modafinil, in combination with cognitive behavior therapy (CBT), to prevent drug relapse among cocaine addicts.

DETAILED DESCRIPTION:
The development of a medication to treat cocaine addiction specifically by lessening withdrawal symptoms has been a primary focus of research. Common cocaine withdrawal symptoms include depression, lack of energy, and poor concentration. Modafinil, a central nervous system stimulant, is a medication that can speed up physical and mental processes in the brain. It is currently used to treat narcolepsy, a condition that causes excessive sleepiness. Modafinil enhances mood, increases energy, and improves concentration in people with narcolepsy. Modafinil may also cause the same effects in individuals addicted to cocaine, thereby countering the symptoms of cocaine withdrawal. The purpose of this study is to compare the effectiveness of modafinil plus CBT versus placebo plus CBT for treating cocaine dependence.

A 2-week screening period will be followed by an 8-week treatment phase. Participants will be randomly assigned to receive either 200 mg of modafinil, 400 mg of modafinil, or placebo on a daily basis for the 8 weeks of treatment. During this time, participants will be asked to report the number of days that they use and do not use cocaine. This will be confirmed three times a week with urine tests. Mood, level of daytime sleepiness, and symptoms of cocaine withdrawal and cocaine "high" will be evaluated. Compliance with study medication will be assessed with urine and blood tests. Medication side effects will be monitored through physical examinations, routine lab tests, ECGs, and self-reports. Follow-up evaluations will occur 4 and 8 weeks following the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Seeking treatment for cocaine dependence
* Meets DSM-IV diagnosis criteria for cocaine dependence as determined by Mini-SCID interview
* If female, willing to use effective contraception throughout the study
* Lives within 50 miles of the research center and has reliable transportation

Exclusion criteria:

* Meets DSM-IV/Mini-SCID diagnosis criteria for dependence on any drugs other than cocaine, alcohol, nicotine, or marijuana
* Physiologic dependence on alcohol requiring medical detoxification, on either an inpatient or outpatient basis
* Current psychiatric disorder, including depression, schizophrenia, bipolar affective disorder, organic brain disease, dementia, or other types of psychosis
* Recent suicidal or homicidal attempts within 60 days of study entry
* Suicidal or homicidal ideation within 30 days of study entry
* Meets diagnosis criteria from the Differential Diagnosis of Psychotic Disorders section of Mini-SCID for a history of psychotic symptoms during a period of cocaine use (e.g., persistent hallucinations and delusions)
* Serious medical illness, including left ventricular hypertrophy, mitral valve prolapse, left bundle branch block, heart attack, angina, serious liver disease (transaminase levels four times greater than normal), and kidney, neurologic, metabolic, neoplastic, nutritional, inflammatory, or endocrine disorders
* Required by the court to obtain treatment for cocaine dependence
* Not seeking treatment for cocaine dependence
* Participated in cocaine treatment (clinical or research) within 30 days of study entry
* Anticipating elective surgery or hospitalization within 20 weeks of study entry
* Known or suspected hypersensitivity to modafinil
* Use of any of the following medications within 14 days of study entry: selective serotonin reuptake inhibitor antidepressants, tricyclic antidepressants, dopamine agonists, and other psychotropic medications, including anticonvulsants, antipsychotics, anxiolytics, or psychostimulants
* Currently taking medications that could adversely interact with study medications, including azole-type antifungals, cyclosporine, warfarin, theophylline, or carbamazepine
* Currently taking any medications that induce or inhibit CYP3A4 metabolic pathways
* Pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2004-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Malcolm, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 200mg Modafinil | 400mg Modafinil | Matching Placebo
Started | 40 | 43 | 40
Completed | 25 | 25 | 17
Not Completed | 15 | 18 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 200mg Modafinil | 400mg Modafinil | Matching Placebo | Total
Number analyzed (Participants) | 40 | 43 | 40 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (7.1) | 40.4 (7.2) | 40.0 (8.8) | 39.8 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 9 | 29
  Male | 30 | 33 | 31 | 94

OUTCOME MEASURES:

1. Primary Outcome: Number of Cocaine Non-use Days
Description: Number of cocaine non-use days was determined by Urine Drug Screen tests which confirmed presence (or no presence) of benzoylecgonine levels.
Time Frame: 8 weeks
Population: The amount of subjects represent those that completed 8 weeks of treatment. The exclusion of alcohol dependence listed in the exclusion criteria within the protocol is referring to a physiological dependence on alcohol requiring a medical detox.
Measure: Mean (Standard Error); unit: Number of Days
Arm/Group | 200mg Modafinil | 400mg Modafinil | Matching Placebo
Number analyzed (Participants) | 25 | 25 | 17
Number of Days
  No Alcohol Dependence: number analyzed (Participants) | 13 | 15 | 9
  No Alcohol Dependence | 10.1 (2.4) | 17.1 (2.3) | 9.3 (2.7)
  Alcohol Dependence: number analyzed (Participants) | 12 | 10 | 8
  Alcohol Dependence | 14.1 (2.5) | 9.4 (2.5) | 12.8 (2.4)

2. Primary Outcome: Percent of Participants With New Use
Description: New Use is defined as a period of at least 7 days abstinence followed by a positive urine drug screen.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 200mg Modafinil | 400mg Modafinil | Matching Placebo
Number analyzed (Participants) | 25 | 25 | 17
Percentage of participants
  No Alcohol Dependence: number analyzed (Participants) | 13 | 15 | 9
  No Alcohol Dependence | 54.2 | 42.0 | 55.8
  Alcohol Dependence: number analyzed (Participants) | 12 | 10 | 8
  Alcohol Dependence | 39.7 | 42.0 | 49.0

ADVERSE EVENTS:
Arm/Group | 200mg Modafinil | 400mg Modafinil | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/43 | 0/40
Other Adverse Events (participants affected / at risk) | 33/40 | 34/43 | 27/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200mg Modafinil (N=40) | 400mg Modafinil (N=43) | Matching Placebo (N=40)
Heart Racing (Cardiac disorders) | 5 (5) | 5 (6) | 1 (1)
Numbness (Nervous system disorders) | 1 (1) | 2 (3) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 13 (17) | 16 (17) | 10 (11)
Muscle Ache (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 7 (7) | 12 (12) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (5) | 8 (8) | 5 (5)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Rapid Heart Rate (Cardiac disorders) | 3 (3) | 3 (3) | 0 (0)
Sleepiness (Psychiatric disorders) | 1 (1) | 2 (3) | 6 (6)
Toothache (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Heartburn (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Chest Pain (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Jitteriness (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes